CLINICAL TRIAL: NCT00943423
Title: A Randomised Phase III Trial to Determine the Role of FDG-PET Imaging in Clinical Stages IA/IIA Hodgkin's Disease
Brief Title: PET Scan in Planning Treatment in Patients Undergoing Combination Chemotherapy For Stage IA or Stage IIA Hodgkin Lymphoma
Acronym: RAPID
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: The Christie NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 03_DOG05_07; CHNT-RAPID; ISRCTN99811594; EU-20931
Record Dates: First submitted 2009-07-20; First posted 2009-07-22 (Estimated); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Lymphoma
Keywords: stage I adult Hodgkin lymphoma; stage II adult Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Active Comparator): Within 6 weeks after completion of course 3 of chemotherapy, patients undergo involved field radiotherapy to disease areas.
  Interventions: Radiation: Involved Field Radiotherapy
- Arm II (Experimental): Patients receive no further treatment.
  Interventions: Other: No further treatment

INTERVENTIONS:
Radiation: Involved Field Radiotherapy — IFRT 30Gy delivered in daily fractions of 1.8 - 2.0Gy
  Arms: Arm I
Other: No further treatment
  Arms: Arm II

SUMMARY:
RATIONALE: A PET scan may help doctors learn how the cancer responded to combination chemotherapy and whether radiation therapy is also required.

PURPOSE: This randomized phase III trial is studying giving a PET scan to see how well it works in deciding whether patients who have received combination chemotherapy for stage IA or stage IIA Hodgkin lymphoma also need radiation therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether patients with stage IA or IIA Hodgkin lymphoma who have a negative fludeoxyglucose F 18 positron emission tomography (FDG-PET) imaging after 3 courses of chemotherapy comprising doxorubicin hydrochloride, bleomycin sulfate, vinblastine, and dacarbazine (ABVD) require consolidation radiotherapy (to areas of previous involvement) in order to delay or prevent disease progression.

OUTLINE: Patients receive doxorubicin hydrochloride IV, bleomycin sulfate IV, vinblastine IV, and dacarbazine IV (ABVD) on days 1 and 15. Treatment repeats every 28 days for 3 courses. On day 15 of the third course of chemotherapy, patients undergo a CT scan of the neck, thorax, abdomen and pelvis. Patients with nonresponsive disease or progressive disease are removed from the study. Patients who achieve response undergo fludeoxyglucose F 18 positron emission tomography (FDG-PET). Patients with a positive FDG-PET scan receive an additional course of ABVD and undergo involved field radiotherapy. Patients with a negative FDG-PET scan are randomized to 1 of 2 treatment arms.

* Arm I: Within 6 weeks after completion of course 3 of chemotherapy, patients undergo involved field radiotherapy to disease areas.
* Arm II: Patients receive no further treatment. After completion of study therapy, patients are followed up every 3 months for 1 year, every 4 months for 1 year, every 6 months for 1 year, and then annually thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed Hodgkin Lymphoma

  * Stage IA or IIA disease

    * No stage IA Hodgkin lymphoma with no clinical or CT evidence of disease after diagnostic biopsy
  * Above the diaphragm with no mediastinal bulk, defined as maximum transverse diameter of mediastinal mass

    * Internal thoracic diameter at level of D5/6 interspace > 0.33
  * Bulky disease at other sites, defined as nodal mass with transverse diameter ≥ 10 cm allowed

PATIENT CHARACTERISTICS:

* Not pregnant or nursing
* Fertile patients must use effective contraception during and for ≥ 6 months
* No prior malignancy except appropriately treated basal cell carcinoma of the skin or carcinoma in situ of the cervix
* No severe underlying illness considered to make the trial therapy hazardous (i.e., severe heart disease or lung fibrosis)
* Willing to travel to the nearest PET scan center
* Able to comply with protocol follow-up arrangements

PRIOR CONCURRENT THERAPY:

* No prior treatment for Hodgkin lymphoma
* No contraindications to chemotherapy or radiotherapy

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 602 (Actual)
Dates: Start 2003-07; Primary Completion 2014-07 (Actual); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | up to 5 years after randomisation

SECONDARY OUTCOMES:
Incidence of FDG-PET scan positivity/negativity after 3 courses of chemotherapy | 3 months after treatment start
Survival and cause of death | up to 5 years after randomisation
Incidence and type of second cancers | up to 5 years after randomisation

CONTACTS AND LOCATIONS:
Overall Officials: John Radford, MD, Principal Investigator — The Christie NHS Foundation Trust
Locations (1):
- Christie Hospital, Manchester, England, United Kingdom

REFERENCES:
- [Derived] Kreuzberger N, Goldkuhle M, von Tresckow B, Kobe C, Sickinger MT, Monsef I, Skoetz N. Positron emission tomography-adapted therapy for first-line treatment in adults with Hodgkin lymphoma. Cochrane Database Syst Rev. 2025 Mar 26;3(3):CD010533. doi: 10.1002/14651858.CD010533.pub3. PMID 40135712
- [Derived] Phillips EH, Counsell N, Illidge T, Andre M, Aurer I, Fiaccadori V, Fortpied C, Neven A, Federico M, Barrington SF, Raemaekers J, Radford J. Maximum tumor diameter is associated with relapse risk in limited-stage Hodgkin lymphoma: an international study. Blood Adv. 2025 May 13;9(9):2266-2274. doi: 10.1182/bloodadvances.2024015140. PMID 39774828
- [Derived] Fiaccadori V, Neven A, Fortpied C, Aurer I, Andre M, Federico M, Counsell N, Phillips EH, Clifton-Hadley L, Barrington SF, Illidge T, Radford J, Raemaekers JMM. Relapse patterns in early-PET negative, limited-stage Hodgkin lymphoma (HL) after ABVD with or without radiotherapy-a joint analysis of EORTC/LYSA/FIL H10 and NCRI RAPID trials. Br J Haematol. 2023 Mar;200(6):731-739. doi: 10.1111/bjh.18594. Epub 2022 Dec 21. PMID 36541117
- [Derived] Cutter DJ, Ramroth J, Diez P, Buckle A, Ntentas G, Popova B, Clifton-Hadley L, Hoskin PJ, Darby SC, Radford J, Illidge T. Predicted Risks of Cardiovascular Disease Following Chemotherapy and Radiotherapy in the UK NCRI RAPID Trial of Positron Emission Tomography-Directed Therapy for Early-Stage Hodgkin Lymphoma. J Clin Oncol. 2021 Nov 10;39(32):3591-3601. doi: 10.1200/JCO.21.00408. Epub 2021 Aug 13. PMID 34388007
- [Derived] Illidge TM, Phillips EH, Counsell N, Pettengell R, Johnson PWM, Culligan DJ, Popova B, Clifton-Hadley L, McMillan A, Hoskin P, Barrington SF, Radford J. Maximum tumor diameter is associated with event-free survival in PET-negative patients with stage I/IIA Hodgkin lymphoma. Blood Adv. 2020 Jan 14;4(1):203-206. doi: 10.1182/bloodadvances.2019001023. PMID 31935289
- [Derived] Barrington SF, Phillips EH, Counsell N, Hancock B, Pettengell R, Johnson P, Townsend W, Culligan D, Popova B, Clifton-Hadley L, McMillan A, Hoskin P, O'Doherty MJ, Illidge T, Radford J. Positron Emission Tomography Score Has Greater Prognostic Significance Than Pretreatment Risk Stratification in Early-Stage Hodgkin Lymphoma in the UK RAPID Study. J Clin Oncol. 2019 Jul 10;37(20):1732-1741. doi: 10.1200/JCO.18.01799. Epub 2019 May 21. PMID 31112475
- [Derived] Radford J, Illidge T, Counsell N, Hancock B, Pettengell R, Johnson P, Wimperis J, Culligan D, Popova B, Smith P, McMillan A, Brownell A, Kruger A, Lister A, Hoskin P, O'Doherty M, Barrington S. Results of a trial of PET-directed therapy for early-stage Hodgkin's lymphoma. N Engl J Med. 2015 Apr 23;372(17):1598-607. doi: 10.1056/NEJMoa1408648. PMID 25901426
- See also: Clinical trial summary from the UCL CTC website — http://www.ctc.ucl.ac.uk/TrialDetails.aspx?Trial=120